CLINICAL TRIAL: NCT03902327
Title: Does N-acetyl-cysteine Treatment Improves Carbohydrate Metabolism in Obese Women?
Brief Title: N-acetyl-cysteine and Carbohydrate Metabolism Disorder in Obese Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Agata Chmurzyńska, dr hab, Director of Institute of Human Nutrition and Dietetics, Poznan University of Life Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PoznanULS
Record Dates: First submitted 2019-03-11; First posted 2019-04-04 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Insulin Resistance; Obesity; Carbohydrate Metabolism Disorder
Keywords: N - acetylocysteine; Obesity; Insulin resistance; Nutrition intervention; Carbohydrate Metabolism
MeSH Terms: conditions — Insulin Resistance; Obesity | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trails
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC group (Experimental): NAC for 12 weeks, 1.6 mg/day, 4x400 mg; a diet based on general recommendations for people with carbohydrate metabolism disorder
  Interventions: Dietary Supplement: NAC group
- Control group (Active Comparator): Placebo for 12 weeks and a diet based on general recommendations for people with carbohydrate metabolism disorder
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: NAC group — Nutrition intervention focused on the treatment of carbohydrate metabolism disorder + N - acetylocysteine supplementation (1600 mg /d, 400 mg x 4 times a day)(30 people).
  Arms: NAC group
Dietary Supplement: Control group — Nutrition intervention focused on the treatment of carbohydrate metabolism disorder + placebo (4 times a day) (30 people).
  Arms: Control group

SUMMARY:
The effect of N-acetylcysteine supplementation on carbohydrate metabolism disorder and homocysteine concentrations in obese women will be analysed.

ELIGIBILITY:
Inclusion criteria:

* women diagnosed with carbohydrate metabolism disorder,
* obesity (BMI >29,9 kg/m2)
* patients not participating in other similar research programs at the same time,
* written agreement to take part in the research.

Exclusion criteria:

* the use of medicament that may affect on carbohydrate metabolism within 4 weeks,
* failure to comply with dietary recommendations established during the nutritional intervention,
* pregnancy and breast feeding.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Insulin Resistance | 12 weeks
  Fasting insulin concentration (uU/ml) will be measured before and after 2 hours of 75g glucose drink. Insulin resistance will be measured before and after 12 weeks of the intervention.
Oral glucose toletance test OGTT | 12 weeks
  Fasting glucose concentration (mg/dL) will be measured before and after 2 hours of 75g glucose drink. OGTT test will be measured before and after 12 weeks of the intervention. Fasting glucose and fasting insulin concentrations will be combined to report HOMA-IR index (homeostatic model assessment of insulin resistance).

SECONDARY OUTCOMES:
Homocysteine concentrations mg/dL | 12 weeks
  Plasma homocysteine concentrations at baseline and after 12 weeks of the intervention
Glutathione level uM/L | 12 weeks
  Plasma glutathione concentrations will be measured at baseline and after 12 weeks of the intervention
Body weight kg | 12 weeks
  Body weight will be assemsment at baseline and after 4,8 and12 weeks of the intervention. Weight and height will be combined to report BMI in kg/m^2.
Body height kg | baseline
  Body height will be assemsment at baseline of the intervention.
Body mass index kg/m2 | 12 weeks
  BMI (body mass index kg/m2) will be assemsment at baseline and after 4, 8 and 12 weeks of the intervention.
Body composition | 12 weeks
  Fat mass (%) and Fat free mass (%) will be assement at baseline and after 4, 8 and 12 weeks of the intervention.
MTHFR polymorphism | baseline
  Methylenetetrahydrofolate reductaseMTHFR polymorphism will be measured only at baseline (before intervention).
Blood lipoproteins measured. | 12 weeks
  Blood lipid profile: cholesterol mg/dL, low-density lipoprotein LDL mg/dL, high-density lipoprotein HDL mg/dL, triglycerides mg/dL will be measured at baseline and after 12 weeks of the intervention.
Cytokine measured | 12 weeks
  Cytokine: IL-6 pg/ml, IL- 10 pg/ml, TNF - α pg/ml will be measured at baseline and after 12 weeks of the intervention.
C-Reactive Protein measured | 12 weeks
  C-Reactive Protein will be measured at baseline and after 12 weeks of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland